CLINICAL TRIAL: NCT04174677
Title: A Phase 2 Open-label, Prospective, Randomized Study of Inebilizumab, VIB4920, or the Combination to Evaluate Safety and Tolerability in Highly Sensitized Candidates Awaiting Kidney Transplantation From a Deceased Donor
Brief Title: Safety and Tolerability of Inebilizumab, VIB4920, or the Combination in Highly Sensitized Candidates Awaiting Kidney Transplantation From a Deceased Donor
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped due to no enrollment
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VIB0551.P2.S1
Record Dates: First submitted 2019-11-05; First posted 2019-11-22 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Highly Sensitized Patients on Waiting List for Kidney Transplantation
Keywords: cPRA, HLA antibodies, kidney transplantation
MeSH Terms: interventions — inebilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Inebilzumab Treatment (Experimental): Infusion of Inebilizumab
  Interventions: Drug: Inebilizumab
- VIB4920 Treatment (Experimental): Infusion of VIB4920
  Interventions: Drug: VIB4920
- Inebilzumab+VIB4920 Treatment (Experimental): Infusion of Inebilizumab and VIB4920
  Interventions: Drug: Inebilzumab+VIB4920

INTERVENTIONS:
Drug: Inebilizumab — Infusion of Inebilizumab
  Arms: Inebilzumab Treatment
Drug: VIB4920 — Infusion of VIB4920
  Arms: VIB4920 Treatment
Drug: Inebilzumab+VIB4920 — Infusion of Inebilizumab and VIB4920
  Arms: Inebilzumab+VIB4920 Treatment

SUMMARY:
Viela Bio is conducting an open-label, randomized study of inebilizumab, VIB4920, or the combination as part of a multi-center study in highly sensitized patients on the deceased donor waiting list for kidney transplantation. Eligible subjects will be randomized to one of three treatment arms, administered the investigational products as an intervention and subsequently followed for safety.

DETAILED DESCRIPTION:
Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with ESRD who are maintained on hemodialysis.
2. Subjects awaiting first or second kidney transplantation from a deceased donor.
3. Subjects with cPRA 98 100% at Screening Visit 1, calculated using antibodies with titer ≥ 1:16 and/or MFI value ≥ 1400, verified by the central laboratory.
4. Subjects with stable anti-HLA antibody titers (a difference of < 2 titers versus the average titer of antibodies compared to the screening sample) based on 2 legacy samples drawn within 6 to 12 months prior to Screening Visit 1, verified by the central laboratory.

Exclusion Criteria:

1. Subjects awaiting kidney transplantation from a living donor.
2. Subjects who have previously undergone desensitization with plasmapheresis/plasma exchange, IVIG, rituximab, imlifidase, tocilizumab or a proteasome inhibitor (eg, bortezomib, carfilzomib, ixazomib, others) within 12 months prior to randomization.
3. Candidates for a second kidney allograft if the first allograft was lost within 12 months prior to screening.
4. Subjects who have experienced a sensitizing event (eg, pregnancy, blood transfusion) within 6 months prior to screening.
5. Recipients of a prior non-kidney organ transplant or stem cell transplant.
6. Subjects treated with systemic immunosuppressive drug therapy for more than a total of 2 weeks within 12 months prior to ICF signature (treatment with corticosteroids < 10 mg/day PO prednisone or equivalent for less than a total of 2 weeks during the 4 weeks prior to screening is allowed).
7. Subjects who have undergone lympho-depleting therapy (eg, Thymoglobulin, alemtuzumab) within 12 months prior to randomization.
8. Subjects with known immunodeficiency.
9. Subjects with known platelet disorders, or history of arterial or venous thromboembolism unrelated to hemodialysis access procedures.
10. Subjects with history of prothrombotic status (including but not limited to congenital or inherited deficiency of antithrombin III, protein C, protein S), or confirmed diagnosis of catastrophic antiphospholipid syndrome.
11. Subjects requiring treatment with antithrombotic drugs (clopidogrel, prasugrel, warfarin, others). Low-dose aspirin treatment (up to 325 mg/day) is allowed.
12. Major surgery within 12 weeks prior to screening.
13. Receipt of live (attenuated) vaccine within the 4 weeks prior to screening.
14. Previous treatment with anti-CD40L agents.
15. Use of B-cell depleting therapy (eg, inebilizumab, rituximab, ocrelizumab, obinutuzumab), non-depleting B-cell directed therapy (eg, belimumab), an anti-CD40 agent, belatacept, or abatacept within 1 year prior to enrollment.
16. Use of anti-interleukin (IL)-6 mAbs (eg, tocilizumab, clazakizumab), C1 esterase inhibitors, or complement inhibitors (eg, eculizumab) or imlifidase within 12 months prior to enrollment.
17. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half lives of enrollment, whichever is longer.
18. Subjects who have had more than one episode of severe infection requiring parenteral antimicrobial treatment within 12 months prior to screening.
19. Subjects with a history of opportunistic infection within 12 months prior to screening (except for PO candidiasis, vaginal candidiasis, and cutaneous fungal infections).
20. Subjects who have had more than one episode of herpes zoster within 12 months prior to screening.
21. Subjects with uncontrolled diabetes mellitus (hemoglobin A1c ≥ 8.0% at screening).
22. Subjects who have a positive test for, or have been treated for, hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection.

    Regarding hepatitis B, positive test for chronic hepatitis B infection at screening, defined as either (1) positive hepatitis B surface antigen (HBsAg) or (2) a positive hepatitis B core antibody (anti-HBcAb)
23. History of or active tuberculosis (TB), or a positive QuantiFERON®-TB Gold test at screening, unless previously treated for latent TB. Subjects with an indeterminate QuantiFERON®-TB Gold test result can repeat the test, but if the repeat test is also indeterminate, they are excluded.
24. History of cancer, except as follows:

    1. In situ carcinoma of the cervix treated with apparent success with curative therapy > 12 months prior to screening; or
    2. Cutaneous basal cell carcinoma treated with apparent success with curative therapy.
25. Any severe cardiovascular, respiratory, endocrine, gastrointestinal, hematological, neurological, psychiatric, or systemic disorder that could impact the evaluation of safety and efficacy assessments or affect the subject's ability to participate in the study or the subject's safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with safety events (treatment-emergent adverse events, treatment-emergent serious adverse events, or treatment-emergent adverse events of special interest) during the course of the study | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Anti-drug antibodies (ADA) of inebilizumab and VIB4920 | Through study completion, an average of 1 year
  The ADA incidence rate will be summarized, where the incidence is the proportion of the subjects with ADA positive post-baseline only or boosted their pre existing ADA during the study period.
Maximum observed concentration of inebilizumab and VIB4920 | Treatment phase of study (Day 1 of treatment to Day 197)
  Pharmacokinetic profile
Area under the concentration-time curve of inebilizumab and VIB4920 | Treatment phase of study (Day 1 of treatment to Day 197)
  Pharmacokinetic profile
Total systemic clearance of inebilizumab and VIB4920 | Treatment phase of study (Day 1 of treatment to Day 197)
  Pharmacokinetic profile

OTHER OUTCOMES:
Proportion of subjects who achieve at least a 1-, 2-, 3-, or 4-titer reduction in anti-HLA antibody strength in at least 25% of antibodies present before treatment versus any post baseline visit | Day 1 through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - Reserach Site California, San Diego, California
  - Pennsylvania Reserach Site, Bethlehem, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing